CLINICAL TRIAL: NCT05238285
Title: Production of Nonverbal Acoustic Signals and Resulting Physiological Responses
Acronym: SINOVE-PRO
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: University of Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 20CH259; 2020-A03457-32: (Other: ANSM)
Record Dates: First submitted 2022-02-02; First posted 2022-02-14 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Self-Perception
Keywords: acoustic analysis; physiological responses; psycho-acoustic tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adult population aged 18 to 80 years: Participants will be asked to produce vocal sounds of different nature according to the non-verbal parameters of interest for the given study.
  Interventions: Behavioral: Production of vocal sounds

INTERVENTIONS:
Behavioral: Production of vocal sounds — Participants will be asked to produce vocal sounds of different nature according to the non-verbal parameters of interest for the given study.
  For example, they can read a script containing vowels ('a', 'e', 'i', 'o', 'u'), short sentences ('hello, how are you'), longer passages of standardised reading texts, and can also be asked to speak freely about any topic ('freedom of speech'). They can be asked to play a role or to imitate a particular emotional state. For example, "imagine that you have just been told that you have won a million euros in the lottery. Produce a vocalisation to express your excitement" or "talk to your dog your dog by imagining that he has done a negative action and then do the same thing by imagining that this time imagining that the action was positive".

SUMMARY:
Like many other animals, humans produce nonverbal vocal signals including screams, grunts, roars, cries and laughter across a variety of contexts. However, despite their importance in the human vocal repertoire, the mechanisms and functions of non-verbal signals remain little studied and poorly understood in humans.Our studies aim to improve our understanding of the nature and function of non-verbal signals.

DETAILED DESCRIPTION:
Like many other animals, humans produce nonverbal vocal signals including screams, grunts, roars, cries and laughter across a variety of contexts. Many of these signals (such as cries) are already produced at birth and likely serve a number of important biological and social functions. In addition, human speech is characterised by nonlinguistic acoustic parameters (such as pitch, formant frequencies, and nonlinear phenomena) that are known to correlate with biologically important traits of the vocalizer.

However, despite their importance in the human vocal repertoire, the mechanisms and functions of non-verbal signals remain little studied and poorly understood in humans.

Theses studies aim to improve the understanding of the nature and function of non-verbal signals. Thus, this study is part of a long-term research project in which investigators are trying to clarify the information contained in the acoustic structure of human non-verbal signals, and to investigate the factors influencing their production.

ELIGIBILITY:
Inclusion Criteria:

- Participant should be affiliated or entitled to a social security scheme

Exclusion Criteria:

* Pregnant women
* Voice production disorders
* Hearing impairment, speech production disorders or major health problems.
* Chronic smoker (more than 10 cigarettes per day)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult population aged 18 to 80 years
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Vocal analysis | During the vocal production
  Participants will receive instructions on what to say or what type of non-verbal vocalisation to produce during the manipulation.
  The vocalisations thus produced by the participants will be systematically recorded and analysed using software adapted to acoustic analysis
  Measurement of acoustic variables such as fundamental frequency (pitch), vocal tract resonances (formants) and vocal disturbances (jitter, shimmer), the nonlinearities and chaotic/noise properties of vocalisations

SECONDARY OUTCOMES:
Heart rate (bpm) | During the vocal production
Skin conductance (Siemens) | During the vocal production
Skin temperature (°C) | During the vocal production
Nociception Level Index (NOL) | During the vocal production
  A non-invasive finger probe, containing four sensors, will be placed on the on the index finger of the participants.
Pupillary diameter (millimeter) | During the vocal production
  Using a high resolution binocular for automated pupil diameter measurement with an infrared camera

CONTACTS AND LOCATIONS:
Overall Officials: ROLAND PEYRON, MDPHD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne; Nicolas MATHEVON, PhD, Study Director — University of Saint-Etienne, France
Locations (1):
- Centre Hospitalier Universitaire de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No